CLINICAL TRIAL: NCT00930007
Title: Comparison of Sleep-wake LH Frequency in Peripubertal Girls With and Without Hyperandrogenemia
Brief Title: Sleep-wake Changes of Luteinizing Hormone Frequency in Pubertal Girls With and Without High Testosterone
Acronym: CRM005
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Virginia (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Chris McCartney, Associate Professor of Medicine, University of Virginia
Other Study IDs: 13950
Record Dates: First submitted 2009-06-24; First posted 2009-06-30 (Estimated); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Hyperandrogenism
Keywords: Luteinizing hormone; Puberty
MeSH Terms: conditions — Hyperandrogenism | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Serum obtained during frequent sampling will be stored (in case repeat measurements are required), but will be discarded at the end of the study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hyperandrogenemic: Girls with elevated free testosterone concentrations
  Interventions: Other: Blood sampling
- Controls: Girls with normal free testosterone concentrations
  Interventions: Other: Blood sampling

INTERVENTIONS:
Other: Blood sampling — Blood sampling for later hormone measurements

SUMMARY:
The purpose of this study is to determine whether sleep-wake changes of luteinizing hormone pulse frequency are different in early pubertal girls with high testosterone levels compared to early pubertal girls with normal testosterone levels.

DETAILED DESCRIPTION:
During early puberty, luteinizing hormone (LH) pulse frequency normally increases during sleep. In contrast, preliminary data suggest that obese girls (who have high testosterone levels in general) demonstrate low LH frequency during the day and night during early puberty; but at mid puberty rapidly transition to a high LH frequency during the day and night. We hypothesize that in early pubertal girls with high testosterone levels, overnight increases of LH frequency are less prominent than those observed in early pubertal girls with normal testosterone levels. We will assess this using a frequent sampling protocol for assessment of LH pulse frequency (with sampling occurring while awake and while asleep) in early pubertal girls with and without high testosterone levels. Sleep will be formally evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Early to midpubertal girls (late Tanner 1 [i.e., estradiol > 20 pg/ml] to Tanner 3)
* Premenarcheal
* Approximate ages, 8-15 years

Exclusion Criteria:

* BMI-for-age < 5th percentile
* Inability to comprehend what will be done during the study or why it will be done
* Being a study of GnRH pulse regulation in adolescent girls with and without HA, boys are excluded
* Obesity associated with a diagnosed (genetic) syndrome (e.g., Prader-Willi syndrome, leptin deficiency), obesity related to medications (e.g., glucocorticoids), etc.
* Pregnancy or lactation
* Virilization
* Total testosterone > 150 ng/dl (confirmed on repeat)
* DHEAS > upper limit of age-appropriate normal range (confirmed on repeat) (mild elevations may be seen in adolescent HA, and elevations < 1.5 times the age-appropriate upper limit of normal will be accepted in such girls)
* Follicular phase 17-hydroxyprogesterone > 250 ng/dl (for girls < 12 years old) or > 300 ng/dl (for girls 12 and older) (confirmed on repeat), which suggests the possibility of congenital adrenal hyperplasia. NOTE: If an elevated follicular 17-hydroxyprogesterone is confirmed on repeat testing, an ACTH stimulated 17-hydroxyprogesterone < 1000 ng/dl will be required for study participation
* History of premature adrenarche (i.e., appearance of pubic and/or axillary hair before age 8)
* A previous diagnosis of diabetes
* Fasting glucose ≥ 126 mg/dl, or a hemoglobin A1c > 6.5% (confirmed on repeat)
* Abnormal TSH (confirmed on repeat) (subjects with adequately treated hypothyroidism, reflected by normal TSH values, will not be excluded)
* Abnormal prolactin (confirmed on repeat) (mild elevations may be seen in HA girls, and elevations < 1.5 times the upper limit of normal will be accepted in this group)
* Evidence of Cushing's syndrome by history or physical exam (e.g., history of impaired growth in children, striae)
* Hematocrit < 36% and hemoglobin < 12 g/dl (confirmed on repeat)
* Significant history of cardiac or pulmonary dysfunction (e.g., known or suspected congestive heart failure; asthma requiring intermittent systemic corticosteroids; etc.)
* Persistent liver test abnormalities (confirmed on repeat), with the exception that mild bilirubin elevations will be accepted in the setting of known Gilbert's syndrome
* Persistently abnormal sodium, potassium, or elevated creatinine concentration (confirmed on repeat)
* Bicarbonate concentrations < 20 or > 30 (confirmed on repeat)
* No medications known to affect the reproductive system, glucose metabolism, lipid metabolism, or blood pressure can be taken in the 3 months prior to the first inpatient GCRC study (or in the 2 months prior to screening)

  * Such medications include oral contraceptive pills, progestins, metformin, glucocorticoids, psychotropics, and sympathomimetics/stimulants (e.g., methylphenidate)
  * Patients taking restricted medications will be excluded unless written permission (for the subjects to discontinue the medication) is received from the subject's physician
* Weight < 22 kg is an absolute exclusion criterion (to ensure safe blood withdrawal)

Ages: 8 Years to 15 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Community sample and patients from local clinics
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2008-10; Primary Completion 2023-05 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Luteinizing hormone pulse frequency (while awake and while asleep) | Baseline (time zero)

SECONDARY OUTCOMES:
Progesterone concentration | Baseline (time zero)
Estradiol concentration | Baseline (time zero)
Testosterone concentrations | Baseline (time zero)
Luteinizing hormone amplitude | Baseline (time zero)
Sleep stage parameters | Baseline (time zero)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher R McCartney, MD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: Undecided
We do not have current plans to share IPD